CLINICAL TRIAL: NCT00454077
Title: Recombinant Human TSH (rhTSH)-Aided Radioiodine (131) Therapy for Thyroid Remnant Ablation in Differentiated Thyroid Cancer Patients: a Comparison Between 1850 MBq and 3700 MBq Activities
Brief Title: rhTSH-Thyroid Ablation With 1850 MBq of 131I
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Other Study IDs: AIRC 1185
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2006-10

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; rhTSH; thyroid ablation
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: radioiodine therapy after rhTSH

SUMMARY:
Most patients with differentiated thyroid carcinoma (DTC) are treated with therapeutic doses of radioiodine (131I) after initial surgery (total or near total thyroidectomy), aimed to destroy microscopic residual normal or tumoral thyroid cells and to facilitate the early detection of tumor recurrence based on serum thyroglobulin (Tg) measurement and 131I whole body scan (WBS) (1-5). Recently, preparation of patients for thyroid ablation with rhTSH and 3700 MBq of 131I on l-thyroxine (l-T4) therapy has been approved in Europe by the European Medicines Agency (EMEA) as an alternative to thyroid hormone withdrawal (6), after a randomized, controlled, multicenter study demonstrated that both methods of preparation are equally effective (with 100% rate of successful ablation) and that patients prepared with rhTSH received lower total body irradiation and experienced a better quality of life compared to those rendered hypothyroid (7).

The present study was aimed to compare the efficacy of fixed activities of 1850 MBq versus 3700 MBq of 131I for post surgical thyroid ablation in DTC patients prepared with rhTSH (TSHα, Thyrogen®, Genzyme Therapeutics, Cambridge, MA) on l-T4 therapy.

DETAILED DESCRIPTION:
Aim: Recently, a multicenter study in differentiated thyroid cancer (DTC) patients showed that 3700 MBq of 131I after rhTSH stimulation had successful post-surgical thyroid ablation rate similar to that obtained after thyroid hormone withdrawal. We investigated whether 1850 MBq of 131I have a rate of successful ablation similar to 3700 MBq in patients prepared with rhTSH.

Methods: Seventy-two patients with DTC were randomly assigned after surgery to receive 1850 MBq (group A, n: 36) or 3700 MBq (group B, n: 36) of 131I after rhTSH. The two groups were comparable for age, sex, histotype and tumor stage. One injection of 0.9 mg of rhTSH was administered for two consecutive days; 131I therapy was delivered 24 hours after the last injection. A post-therapy whole body scan (WBS) was performed 72 hours later. Successful ablation was assessed 6-8 months after therapy.

Results: Successful ablation, defined as no visible uptake in the diagnostic WBS after rhTSH stimulation, was achieved in 88.9% of group A and group B patients. Basal and rhTSH-stimulated serum Tg was undetectable (<1 ng/ml) in 88.6 % of group A and 84.8% of group B patients (p=0.65). Similar rates of ablation were obtained in both groups also in patients with lymph node metastases. Dosimetric data showed similar thyroid bed uptake, effective half-life and adsorbed dose in the two groups. Failure to ablate was not correlated with TNM staging, peak TSH levels, thyroid bed uptake and urinary iodine excretion at the time of ablation, but was influenced by the absorbed dose of 131I (< or >300 Gy).

Conclusion: Our results demonstrate that therapeutic 131I activities of 1850 MBq are equally effective as 3700 MBq for thyroid ablation in DTC patients prepared with rhTSH, even in the presence of lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed differentiated thyroid cancer patients, more than 18 years old, recently treated by near total thyroidectomy were eligible for the study

Exclusion Criteria:

* Evidence of distant metastases and/or significant local invasion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2004-12; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Furio Pacini, MD, Principal Investigator — Section of Endocrinology, University of Siena
Locations (1):
- Section of Endcrinology, University of Siena, Siena, Siena, Italy